CLINICAL TRIAL: NCT03412435
Title: Asan Medical Center Myocardial Infarction Registry
Acronym: Asan-MI
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Cardiology, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2018-01
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Myocardial Infarction, Acute; Coronary Stenosis
Keywords: Acute myocardial infarction; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myocardial infarction: diagnosed as acute myocardial infarction and treated with medical treatment, coronary artery bypass surgery and percutaneous coronary intervention.

SUMMARY:
This study evaluates long-term outcome of patients diagnosed as acute myocardial infarction and treated with medication, coronary artery bypass surgery and percutaneous coronary intervention in Asan medical center, Korea.

DETAILED DESCRIPTION:
This study will collect 3000 cases retrospectively and 2000 cases prospectively.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive acute myocardial infarction patients diagnosed through coronary angiography

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive acute myocardial infarction patients diagnosed through coronary angiography
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-04-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
A composite event of all-cause death, non-fatal myocardial infarction and repeat revascularization | 1 year

SECONDARY OUTCOMES:
All cause death | 5 year
Cardiac death | 5 year
Myocardial infarction | 5 year
A composite event of all-cause death and myocardial infarction | 5 year
A composite event of cardiac death and myocardial infarction | 5 year
Repeat revascularization | 5 year
Stent thrombosis | 5 year
  according to Academic Research Consortium (ARC) criteria
Stroke | 5 year
  A stroke or cerebrovascular accident with loss of neurological function caused by an ischemic or hemorrhagic event with residual symptoms at least 24 hours after onset or leading to death.
Procedure success | 7 days
  Successful percutaneous coronary intervention at the intended target lesion with final instant residual stenosis of less than 30% by quantitative coronary angiography (QCA) and no event of death or Q wave myocardial infarction or urgent revascularization during hospitalization.
Surgery success | 7 days
  Successful surgery defines as no event of death or Q wave myocardial infarction or urgent revascularization during hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided